CLINICAL TRIAL: NCT03098953
Title: Evaluation of the Safety, Systemic Pharmacokinetics, and Tolerability of Single and Repeat Ocular Instillations of LE Ophthalmic Gel
Brief Title: Evaluation of the Safety, Systemic Pharmacokinetics, and Tolerability of Single and Repeat Ocular Installations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 881
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Ocular Installation
MeSH Terms: interventions — Loteprednol Etabonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Loteprednol Etabonate Ophthalmic Gel (Experimental): one drop per eye for each eye
  Interventions: Drug: Loteprednol Etabonate

INTERVENTIONS:
Drug: Loteprednol Etabonate — one drop per eye for each eye
  Other Names: LE gel

SUMMARY:
Evaluation of the Safety, Systemic Pharmacokinetics, and Tolerability of Single and Repeat Ocular Instillations of Loteprednol Etabonate Ophthalmic Gel

DETAILED DESCRIPTION:
This will be a single-center, single-arm, open label PK clinical study of loteprednol etabonate (LE) ophthalmic gel, 0.38% conducted at one clinical center in the United States (US), with the goal of enrolling approximately 15 healthy normal subjects in the treatment period

ELIGIBILITY:
Inclusion Criteria:

1. Are able to read, understand and provide written informed consent on an Informed Consent Form (ICF) approved by the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
2. Be a non-smoking male or female at least 18 years of age on the date the ICF is signed and with the capacity to provide voluntary informed consent.
3. Be in general good health and free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or place the subject at increased risk during the study.
4. Be willing/able to return for all required study visits and follow instructions from the study Investigator and his/her staff.
5. Are able to self-administer eye drops or have a clinical staff member deliver the single dose of investigational product (IP) on specified study days.

Exclusion Criteria:

1. Have a history/presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject, confound the result(s) of the study, or preclude study treatment or follow-up.
2. Have any current disease or medical condition that requires medicinal therapy.
3. Have a history of drug or alcohol abuse in the last 6 months.
4. Have a positive urine screen for alcohol, amphetamines, barbiturates, benzodiazepines, cocaine (or cocaine metabolite), cannabinoids, methadone, methamphetamine, opiates and/or phencyclidine.
5. Are known to have a prior positive blood screen for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus types 1 and 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
PK analysis will be performed using standard non compartmental method | Day15/Day1
  When possible, plasma concentrations by scheduled time point and PK parameters (AUC0-t (Area under the time-concentration curve to the last measured time point) will be summarized using descriptive statistics by Visit.
PK analysis will be performed using standard non compartmental method | Day 15/Day 1
  When possible, plasma concentrations by scheduled time point and PK parameters, AUC0-∞(Area under the time-concentration curve extrapolated to infinity) will be summarized using descriptive statistics by Visit.
PK analysis will be performed using standard non compartmental method | Day15/Day1
  When possible, plasma concentrations by scheduled time point and PK parameters Cmin (Minimum drug plasma concentration) will be summarized using descriptive statistics by Visit.
PK analysis will be performed using standard non compartmental method | Day15/Day1
  When possible, plasma concentrations by scheduled time point and PK parameters Cmax (Maximum drug plasma concentration), Cmin (Minimum drug plasma concentration) will be summarized using descriptive statistics by Visit.
PK analysis will be performed using standard non compartmental method | Day15/Day1
  When possible, plasma concentrations by scheduled time point and PK parameters RAUC (Ratio (Visit 3/Visit 2) for AUC0-t) will be summarized using descriptive statistics by Visit.
PK analysis will be performed using standard non compartmental method | Day15/Day1
  When possible, plasma concentrations by scheduled time point and PK parameters RCmax (Ratio (Visit 3/Visit 2) for Cmax) will be summarized using descriptive statistics by Visit.
PK analysis will be performed using standard non compartmental method | Day15/Day1
  When possible, plasma concentrations by scheduled time point and PK parameters Tmax (Time at which maximum plasma concentration achieved) will be summarized using descriptive statistics by Visit.
PK analysis will be performed using standard non compartmental method | Day15/Day1
  When possible, plasma concentrations by scheduled time point and PK parameters Kel (Elimination rate constant) will be summarized using descriptive statistics by Visit.
PK analysis will be performed using standard non compartmental method | Day 15/Day 1
  When possible, plasma concentrations by scheduled time point and PK parameters T1/2 (Plasma drug concentration half-life)) will be summarized using descriptive statistics by Visit

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Valeant Site 01, Inglewood, California, United States

IPD SHARING:
Plan to Share IPD: Yes